CLINICAL TRIAL: NCT07401251
Title: Lead Exposure Intervention Program
Acronym: LEIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Sarah Benki-Nugent, Associate Professor, Department of Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00022114; 1R01ES036010 (NIH)
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lead Exposure; High Blood Lead Levels
Keywords: lead; pediatric; Sub-Saharan Africa; lead risk reduction
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate messages (Active Comparator): Caregivers of children with elevated blood lead levels will be provided with immediate messages about lead risk mitigation in the clinic setting. They will receive follow-up at 3 months and 9 months and will complete recall, behavior, and recheck questionnaires and their children will have BLL rechecks.
  Interventions: Behavioral: In-clinic lead risk reduction intervention
- Home visit (Experimental): Caregivers of children with elevated blood lead levels will be provided with immediate messages about lead risk mitigation in the clinic setting. They will also receive a home observation visit and have those risk reduction methods reiterated and tailored to their home situation. They will receive follow-up at 3 months and 9 months and will complete recall, behavior, and recheck questionnaires and their children will have BLL rechecks.
  Interventions: Behavioral: Home visit with tailored messages; Behavioral: In-clinic lead risk reduction intervention

INTERVENTIONS:
Behavioral: Home visit with tailored messages — The home visit will be conducted within 2 weeks of initial screening. During the home visit, the lead exposure risk survey will be re-administered, for comparison to in-clinic self-report survey responses. In addition, an observational checklist of potential lead exposure risk factors will be conducted to identify and discuss residential features and items in the home environment that may be influencing their BLL. Tailored messages on lead exposure risk reduction will be provided.
  A random sample of caregivers will complete an in-depth interview to gather barriers, understandability, and acceptability of the lead risk reduction messages received.
  Arms: Home visit
Behavioral: In-clinic lead risk reduction intervention — For children with BLL < 5 ug/dL, the result will be provided to the caregiver, together with standard post-test messaging on reducing lead exposure. A job-aid, such as a poster, showing common sources of lead exposure in children, and important sources of iron rich foods will be used to guide messaging. For BLLs ≥ 5, tailored messaging on potential sources identified on the risk factor survey will be provided.
  A random sample of caregivers will complete an in-depth interview to gather barriers, understandability, and acceptability of the lead risk reduction messages received.

SUMMARY:
The goal of this clinical trial is to learn if BLL (blood lead level) screening and "healthy home" lead prevention program created in the US is adaptable to a Sub-Saharan African context. It will also work to address child lead exposure in Nairobi, Kenya. The main questions it aims to answer is:

* Can materials and protocols developed for a US audience be effective in a Sub-Saharan African one?
* Is there a difference in learning and action between groups that receive different degrees of intervention?

Researchers will compare the outcomes of a group that received lead risk reduction information only in the clinical setting to a group that also received a home visit and tailored risk reduction messages.

Participants will:

* Have their child's blood lead levels measured at several timepoints
* Take part in a questionnaire about lead risk
* Receive lead risk reduction messaging either only in the clinic setting or also in their homes
* Have their knowledge and risk reduction behaviors measured

ELIGIBILITY:
Inclusion Criteria:

* Caregivers with children ages 12-72 months attending routine care/vaccination visit at Nairobi clinical site.

Exclusion Criteria: Children outside of age range, caregivers younger than 18; plan to leave study catchment within 9 months.

-

Ages: 12 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Recall of survey risk factors | 3 and 9 months post clinic visit
  Lead risk surveys will be completed by participants during the clinic visit and at 3 and 9 months post home visit. Qualitative analysis of the lead risk survey will summarize themes on understandability and acceptability of survey items and messages. The rapid analysis will also explore facilitators and barriers to uptake of recommended exposure reduction measures, and individual level determinants associated with uptake (e.g., empowerment, self-efficacy).
Self report of risk-reduction behavior | 3 and 9 months post clinic visit
  Assess the proportion of caregivers self-reporting uptake of at least one of their risk reduction recommendations within arms and by BLL.

SECONDARY OUTCOMES:
Differences in outcomes between arms | 3 and 9 months post clinic visit
  Using risk survey responses and self-reported changes in risk reduction behavior, we will compare the participants of both arms to assess for differences.

OTHER OUTCOMES:
Uptake of the BLL re-check | 3 and 9 months post-initial visit
  Return for a re-check visit is an indicator of caregiver awareness of importance of reducing lead exposure. We will summarize the proportions of caregivers returning for each BLL re-check visit for each arm.
Change in BLL | 3 and 9 months post-initial clinic visit
  Change in BLL at re-checks. We do not anticipate observing a significant reduction in child BLL, given that caregivers might not have the ability to identify and/or modify a lead risk exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Benki-Nugent, Principal Investigator — University of Washington
Locations (1):
- Pumwani Hospital and Baba Ndogo Health Centre, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All data other than patient direct or indirect identifiers will be shared.
Access Criteria: Other researchers can contact the MPIs and complete an approved Data Sharing Agreement